## "Poised for Parkinson's"

Informed Consent for Participation in a Study of Online Alexander Technique Classes for People Living with Parkinson's Disease and their Care Partners

Contact information for this study:
Monika Gross, Executive Director of the Poise Project
828-254-3102 monika.gross@thepoiseproject.org

Document Date: May 24, 2021

ClinicalTrials.gov NCT04726709

Principal Investigator: Rajal G. Cohen, rcohen@uidaho.edu

## "Poised for Parkinson's"

## Informed Consent for Participation in a Study of Online Alexander Technique Classes for People Living with Parkinson's Disease and their Care Partners

- 1. This study has been approved by the Institutional Review Board of the University of Idaho.
- 2. **The purpose of this study** is to find out whether people living with Parkinson's disease and their care partners will benefit from online Alexander technique group classes in the management of their daily physical and emotional challenges. We hope to use this information to understand how online Alexander technique classes can be a strategy for improving the lives of people living with Parkinson's. Alexander technique is an educational approach that teaches self-awareness skills for managing the physical and emotional demands of daily life.
- 3. You will benefit directly from this study by receiving online Alexander classes at no cost. We hope that other people living with Parkinson's disease and their care partners will benefit from the inclusion of your shared data and experiences by allowing us to improve our online classes and to increase the possibility for funding for future online classes to be made available to other people living with Parkinson's and their care partners.
- 4. Before the classes begin and after all the classes are over you will complete **surveys** about how you experience the physical and emotional challenges of living with Parkinson's. The estimated time to complete each survey session is no more than 30 minutes.
- 5. You will be given an **evaluation form** about your experience after all the classes are over. The estimated time to complete this form is no more than 15 minutes.
- 6. People living with Parkinson's who are participants will also be scheduled for two individual online **physical assessment sessions**, one before the classes begin and one after all the classes are over. At these 60 minute sessions, a researcher will help conduct some assessments including some **videos** taken of you doing simple activities such as sitting, standing and walking. Your care partner will be helping you during this online assessment.
- 7. You may possibly also be contacted after 3 months and 6 months and scheduled to repeat the **follow up surveys** that you originally did.
- 8. There is always a possibility that you may experience embarrassment or anxiety before, during, or after your participation in any classes. As in any normal class involving movement, you may slip, trip, lose your balance, feel physically tired, or fall during participation. We estimate from past experience that these things are not any more likely to happen in our classes than in your normal everyday life. Your comfort and safety is important to us; both your class instructor and the person administering the surveys and measures will do their best to protect you from any risk of injury and distress.

- 9. You are free to stop participation in this study at any time. If you decide to stop participation, all you have to do is tell the Alexander teacher or study coordinator that you no longer wish to participate. You may also chose at any time not to participate in a particular activity or interaction of any class, or of any survey or research component, while still being able to chose to continue to participate in other parts.
- 10. Your participation in this study will be kept confidential. Participant IDs and data (including video records) will be kept in a separate location from the list of participant names, and only those researchers involved in this study will have access to this information. In any poster or photo or text of this study, you will be identified simply as "Participant #1" or "Participant #2" and so forth.
- 11. If you have any questions now or later, we will answer them to the best of our ability.
- 12. Contact information for this study:

Monika Gross, Executive Director of the Poise Project 828-254-3102 monika.gross@thepoiseproject.org

Yes, please blur my facial features

I am 18 years old or older and have reviewed this consent form and understand and agree to its contents.

| Name of Participant | Signature | Date |
|---|---|---|
| Name of Researcher | Signature | Date |
| Please initial any or all of the follo | owing lines regarding use of images: | |
| I grant permission for unidentified is scientific publications or conference | mages or video recordings of me collectes. | eted during this study to be used for |
| I grant permission for unidentified in other educational purposes in print | images or video recordings of me collector online. | eted during this study to be used for |
| If you initialed the second line ab | ove, please select one of the two optio | ns below: |
| Would you like your facial features public? | to be blurred in any research photos or | video images that are viewed by the |
| No, blurring my facial featu | res is not necessary | |